CLINICAL TRIAL: NCT07076966
Title: Comparison of the Performance Between Conventional Colonoscopy and 3D Colonoscopy in Surveillance Colonoscopy: A Multi-center, Randomized Controlled Trial
Brief Title: Comparison of Adenoma Detection Rate in 3D vs. 2D Surveillance Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Attending physician, Department of Internal Medicine, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 202311019DIPC
Record Dates: First submitted 2024-10-22; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Colonoscopy; Adenoma Detection Rate; Three Dimensional; Colon Polyps and Adenomas
Keywords: Colonoscopy; adenoma detection rate; 3D; surveillance colonoscopy
MeSH Terms: conditions — Colonic Polyps; Adenoma

STUDY DESIGN:
Intervention Model Description: 3D colonoscopy versus standard 2D colonoscopy
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D colonoscopy (Experimental)
  Interventions: Device: 3D device
- 2D colonoscopy (No Intervention)

INTERVENTIONS:
Device: 3D device — Use 3D machine to generate the 3D image
  Arms: 3D colonoscopy

SUMMARY:
There is substantial evidence confirming that identifying and removing colorectal adenomas during colonoscopy helps prevent the development of colorectal cancer. Among the quality indicators for colonoscopy, adenoma detection rate (ADR) is the most important, as it is closely related to the patient's future risk of colorectal cancer. Recent studies have further demonstrated that improving ADR can reduce future mortality from colorectal cancer. Notably, non-polypoid lesions (such as flat or depressed lesions) are more likely to be missed during traditional colonoscopy, making these lesions a leading cause of post-colonoscopy interval colorectal cancer.

In a prospective trial conducted by our team comparing the ADR of 3D colonoscopy with standard 2D colonoscopy, we found that 3D colonoscopy significantly improved overall ADR and the detection rate of non-polypoid adenomas.

According to current international guidelines, after an index colonoscopy, patients are recommended to undergo surveillance colonoscopy 1 to 10 years later, depending on their findings at index colonoscopy. Since these patients represent the majority in clinical practice, increasing the ADR during surveillance colonoscopy not only allows for more precise recommendations for the timing of the next colonoscopy but also effectively reduces the risk of post-colonoscopy colorectal cancer (PCCRC).

Therefore, this multicenter, prospective, randomized trial aims to compare the clinical performance of 3D colonoscopy and standard 2D colonoscopy in the context of surveillance colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 40 years of older
* Subjects who receive colonoscopy and polypectomy more the 1 year
* Subjects who need surveillance colonoscopy

Exclusion Criteria:

* Contraindication for colonoscopy
* Subjects with familiar or hereditary polyposis
* Subjects with history of colectomy
* Inadequate bowel cleansing level
* Subjects with inflammatory bowel disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 30 minutes

SECONDARY OUTCOMES:
Flat-ADR | 30 minutes
  detection rate of flat adenoma
Proximal ADR | 30 minutes
  detection rate of adenoma at proximal colon
Distal ADR | 30 minutes
  detection rate of adenoma at distal colon
SSLDR | 30 minutes
  detection rate of sessile serrated lesion
AADR | 30 minutes
  detection rate of advanced adenoma
Detection of of adenoma with various size | 30 minutes
Polyp detection rate | 30 minutes
Adenoma number per colonoscopy, | 30 minutes
Polyp number per colonoscopy | 30 minutes

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Hsinchu Branch, Hsinchu, Taiwan
  - National Taiwan University Cancer Center, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan